CLINICAL TRIAL: NCT05832918
Title: Effects of Core Stability Exercises and Cognitive Tasks Compared to General Exercises and Cognitive Tasks on Chronic Non-specific Back Pain
Brief Title: Effects of Core Stability Exercises and Cognitive Tasks on Chronic Non-specific Back Pain
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Reza Salehi, Iran University of Medical Sciences, Iran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IUMS
Record Dates: First submitted 2023-03-31; First posted 2023-04-27 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Chronic Non-specific Low Back Pain
Keywords: Low back pain; Disability; Postural control; Core Stability Exercise; cognitive task
MeSH Terms: conditions — Low Back Pain | interventions — Exercise Therapy

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- core stability exercises with cognitive tasks group (Experimental): This research will use core stability exercises to strengthen local muscles (transversus abdominis and multifidus) based on the training program provided by Shamsi et al., which is modified from the exercise program of Koumantakis et al.. Participants will be treated for six weeks, three sessions a week, and 16 sessions.
  We will also combine stabilization exercises with cognitive tasks.
  Interventions: Other: exercise therapy
- general exercises with cognitive tasks group (Active Comparator): This research will use general exercises to strengthen global muscles (abdominal flexor muscles and back extensor muscles) based on the training program provided by Shamsi et al.(110), which is modified by Koumantakis et al.. Participants will be treated for six weeks, three sessions a week, and 16 sessions.
  We will also combine general exercises with cognitive tasks.
  Interventions: Other: exercise therapy

INTERVENTIONS:
Other: exercise therapy — Exercise therapy is one of the rehabilitation methods that is defined as a regimen or plan of physical activities designed and prescribed to facilitate the patient's recovery from diseases and any conditions which disturb their movement and activity of daily life or maintain a state of well-being through neuro re-education, gait training, and therapeutic exercises.

SUMMARY:
This randomized control trial study aims to compare the effect of core stability exercises and cognitive tasks with general exercises and cognitive tasks on pain, disability, and postural control strategies of chronic non-specific low back pain patients. The main questions are:

1. Are core stability exercises and cognitive tasks more effective than general exercises and cognitive tasks in reducing the pain of chronic non-specific low back pain patients?
2. Are core stability exercises and cognitive tasks more effective than general exercises and cognitive tasks in reducing the disability of chronic non-specific low back pain patients?
3. Are core stability exercises and cognitive tasks more effective than general exercises and cognitive tasks in improving postural stability parameters of chronic non-specific low back pain patients?
4. Are core stability exercises and cognitive tasks more effective than general exercises and cognitive tasks in improving stabilogram diffusion analysis parameters of chronic non-specific low back pain patients? This study is designed to apply two exercise protocols on two groups of 17 people with non-specific back pain. Group A will receive core stability exercises along with cognitive tasks, and group B will receive general exercises along with cognitive tasks.

DETAILED DESCRIPTION:
Patients will be aged between 18-50 years. All patients meeting the inclusion criteria will receive 16 training sessions (thrice a week). The primary outcome measure will be pain and disability. Secondary outcome measures will be postural control strategies (including postural control stability and stabilogram diffusion analysis), quality of life, fear of movement, and fear-avoidance beliefs that will be assessed before and after training sessions and at 3-month follow-up; only primary outcomes will be evaluated in each group.

ELIGIBILITY:
Inclusion Criteria:

* Orthopedist-confirmed diagnosis of chronic nonspecific low back pain that has lasted at least three months since its onset.
* Pain score of 3 or more on a visual analog scale.
* Pain during quiet standing.
* Cognitive level above 24 based on mini-mental state examination (MMSE).

Exclusion Criteria:

* Radicular pain and any neurological signs.
* Uncorrected vision impairment.
* Hearing problems.
* Vestibular dysfunctions.
* Cognitive deficit.
* Previous spinal surgery.
* Severe deformity or injury to the lower extremities.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 48 (Estimated)
Dates: Start 2023-05-02 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-15 (Estimated)

PRIMARY OUTCOMES:
Oswestry Disability Index | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks ", "change from baseline at three months "
  Questionnaire evaluating the level of disability. Total score range from 0-100 (higher scores mean more disability)

SECONDARY OUTCOMES:
Center of pressure (COP) sway range for anteroposterior (AP range) | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  AP range is one kind of COP displacement evaluation method characterized as traditional linear measures for evaluating postural control stability.
COP sway range for mediolateral (MA range) | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  MA range is one kind of COP displacement evaluation method characterized as traditional linear measures for evaluating postural control stability.
COP sway velocity | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  COP sway velocity is one kind of COP displacement evaluation method characterized as traditional linear measures for evaluating postural control stability.
Sway area | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  Sway area is one kind of COP displacement evaluation method characterized as traditional linear measures for evaluating postural control stability.
Short-term diffusion coefficient of stabilogram diffusion plot | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  The short-term diffusion coefficient is the slope of the open-loop part of the stabilogram diffusion plot, indicating stochastic activity in open loop control phase in a quiet standing position.
Long-term diffusion coefficient of stabilogram diffusion plot | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  The long-term diffusion coefficient is the slope of the close loop part of the stabilogram diffusion plot, indicating stochastic activity in the immediate loop control phase in the quiet standing position.
Critical point coordinates. | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  Critical point coordinates are the estimated values of the time intervals and mean square displacements defining the stabilogram-diffusion critical points (the point that open-loop control changed to close loop control)
12-item short form health survey | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  Questionnaire evaluating the quality of life. Total score range from 0-100 (higher scores mean better quality of life)
Tampa scale for kinesiophobia | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  Questionnaire evaluating the kinesiophobia because of feeling re-injury. Total score range from 17-68 (higher scores mean more kinesiophobia)
Fear-avoidance beliefs questionnaire | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks "
  Questionnaire evaluating fear of pain and consequent avoidance of physical activity because of their fear. Total score range from 0-66 (higher scores mean more fear of pain)
Visual analog scale | "Baseline (pre-intervention)", "change from baseline immediately after the intervention at five weeks ", "change from baseline at three months "
  Questionnaire evaluating pain intensity. Total score range from 0-10 (higher scores mean more pain)

CONTACTS AND LOCATIONS:
Overall Officials: Zeinab Raoufi, PhD student, Principal Investigator — Department of Physiotherapy, School of Rehabilitation Sciences, Iran University of Medical Sciences; Reza Salehi, PhD, Study Director — Department of Physiotherapy, School of Rehabilitation Sciences, Iran University of Medical Sciences
Locations (1):
- Iran University of Medical Sciences, Tehran, Iran (the Islamic Republic Of), Iran

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Frizziero A, Pellizzon G, Vittadini F, Bigliardi D, Costantino C. Efficacy of Core Stability in Non-Specific Chronic Low Back Pain. J Funct Morphol Kinesiol. 2021 Apr 22;6(2):37. doi: 10.3390/jfmk6020037. PMID 33922389
- [Background] Agnus Tom A, Rajkumar E, John R, Joshua George A. Determinants of quality of life in individuals with chronic low back pain: a systematic review. Health Psychol Behav Med. 2022 Jan 5;10(1):124-144. doi: 10.1080/21642850.2021.2022487. eCollection 2022. PMID 35003902
- [Background] van Tulder M, Becker A, Bekkering T, Breen A, del Real MT, Hutchinson A, Koes B, Laerum E, Malmivaara A; COST B13 Working Group on Guidelines for the Management of Acute Low Back Pain in Primary Care. Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care. Eur Spine J. 2006 Mar;15 Suppl 2(Suppl 2):S169-91. doi: 10.1007/s00586-006-1071-2. No abstract available. PMID 16550447
- [Background] Lamoth CJ, Stins JF, Pont M, Kerckhoff F, Beek PJ. Effects of attention on the control of locomotion in individuals with chronic low back pain. J Neuroeng Rehabil. 2008 Apr 25;5:13. doi: 10.1186/1743-0003-5-13. PMID 18439264
- [Background] Kanekar N, Aruin AS. Aging and balance control in response to external perturbations: role of anticipatory and compensatory postural mechanisms. Age (Dordr). 2014 Jun;36(3):9621. doi: 10.1007/s11357-014-9621-8. Epub 2014 Feb 16. PMID 24532389
- [Background] Hodges PW, Richardson CA. Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis. Spine (Phila Pa 1976). 1996 Nov 15;21(22):2640-50. doi: 10.1097/00007632-199611150-00014. PMID 8961451
- [Background] Bussey MD, Aldabe D, Shemmell J, Jowett T. Anticipatory postural control differs between low back pain and pelvic girdle pain patients in the absence of visual feedback. Hum Mov Sci. 2020 Feb;69:102529. doi: 10.1016/j.humov.2019.102529. Epub 2019 Nov 11. PMID 31726292
- [Background] Hodges PW. Changes in motor planning of feedforward postural responses of the trunk muscles in low back pain. Exp Brain Res. 2001 Nov;141(2):261-6. doi: 10.1007/s002210100873. PMID 11713638
- [Background] Mitchell SL, Collins JJ, De Luca CJ, Burrows A, Lipsitz LA. Open-loop and closed-loop postural control mechanisms in Parkinson's disease: increased mediolateral activity during quiet standing. Neurosci Lett. 1995 Sep 8;197(2):133-6. doi: 10.1016/0304-3940(95)11924-l. PMID 8552278
- [Background] Collins JJ, De Luca CJ. Open-loop and closed-loop control of posture: a random-walk analysis of center-of-pressure trajectories. Exp Brain Res. 1993;95(2):308-18. doi: 10.1007/BF00229788. PMID 8224055
- [Background] Collins JJ, De Luca CJ, Burrows A, Lipsitz LA. Age-related changes in open-loop and closed-loop postural control mechanisms. Exp Brain Res. 1995;104(3):480-92. doi: 10.1007/BF00231982. PMID 7589299
- [Background] Wong JJ, Cote P, Sutton DA, Randhawa K, Yu H, Varatharajan S, Goldgrub R, Nordin M, Gross DP, Shearer HM, Carroll LJ, Stern PJ, Ameis A, Southerst D, Mior S, Stupar M, Varatharajan T, Taylor-Vaisey A. Clinical practice guidelines for the noninvasive management of low back pain: A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration. Eur J Pain. 2017 Feb;21(2):201-216. doi: 10.1002/ejp.931. Epub 2016 Oct 6. PMID 27712027
- [Background] Owen PJ, Miller CT, Mundell NL, Verswijveren SJJM, Tagliaferri SD, Brisby H, Bowe SJ, Belavy DL. Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis. Br J Sports Med. 2020 Nov;54(21):1279-1287. doi: 10.1136/bjsports-2019-100886. Epub 2019 Oct 30. PMID 31666220
- [Background] Koumantakis GA, Watson PJ, Oldham JA. Trunk muscle stabilization training plus general exercise versus general exercise only: randomized controlled trial of patients with recurrent low back pain. Phys Ther. 2005 Mar;85(3):209-25. PMID 15733046
- [Background] Hlaing SS, Puntumetakul R, Khine EE, Boucaut R. Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial. BMC Musculoskelet Disord. 2021 Nov 30;22(1):998. doi: 10.1186/s12891-021-04858-6. PMID 34847915
- [Background] Coulombe BJ, Games KE, Neil ER, Eberman LE. Core Stability Exercise Versus General Exercise for Chronic Low Back Pain. J Athl Train. 2017 Jan;52(1):71-72. doi: 10.4085/1062-6050-51.11.16. Epub 2016 Nov 16. PMID 27849389
- [Background] Saragiotto BT, Maher CG, Yamato TP, Costa LOP, Costa LCM, Ostelo RWJG, Macedo LG. Motor Control Exercise for Nonspecific Low Back Pain: A Cochrane Review. Spine (Phila Pa 1976). 2016 Aug 15;41(16):1284-1295. doi: 10.1097/BRS.0000000000001645. PMID 27128390
- [Background] Ganesh GS, Kaur P, Meena S. Systematic reviews evaluating the effectiveness of motor control exercises in patients with non-specific low back pain do not consider its principles - A review. J Bodyw Mov Ther. 2021 Apr;26:374-393. doi: 10.1016/j.jbmt.2020.08.010. Epub 2020 Sep 6. PMID 33992272
- [Background] Remy F, Wenderoth N, Lipkens K, Swinnen SP. Dual-task interference during initial learning of a new motor task results from competition for the same brain areas. Neuropsychologia. 2010 Jul;48(9):2517-27. doi: 10.1016/j.neuropsychologia.2010.04.026. Epub 2010 Apr 29. PMID 20434467
- [Background] Burcal CJ, Needle AR, Custer L, Rosen AB. The Effects of Cognitive Loading on Motor Behavior in Injured Individuals: A Systematic Review. Sports Med. 2019 Aug;49(8):1233-1253. doi: 10.1007/s40279-019-01116-7. PMID 31066022
- [Background] Hemmati L, Piroozi S, Rojhani-Shirazi Z. Effect of dual tasking on anticipatory and compensatory postural adjustments in response to external perturbations in individuals with nonspecific chronic low back pain: Electromyographic analysis. J Back Musculoskelet Rehabil. 2018;31(3):489-497. doi: 10.3233/BMR-170992. PMID 29332033
- [Background] Wang XQ, Zheng JJ, Yu ZW, Bi X, Lou SJ, Liu J, Cai B, Hua YH, Wu M, Wei ML, Shen HM, Chen Y, Pan YJ, Xu GH, Chen PJ. A meta-analysis of core stability exercise versus general exercise for chronic low back pain. PLoS One. 2012;7(12):e52082. doi: 10.1371/journal.pone.0052082. Epub 2012 Dec 17. PMID 23284879
- [Background] Woollacott M, Shumway-Cook A. Attention and the control of posture and gait: a review of an emerging area of research. Gait Posture. 2002 Aug;16(1):1-14. doi: 10.1016/s0966-6362(01)00156-4. PMID 12127181
- [Background] Sherafat S, Salavati M, Takamjani IE, Akhbari B, Rad SM, Mazaheri M, Negahben H, Lali P. Effect of dual-tasking on dynamic postural control in individuals with and without nonspecific low back pain. J Manipulative Physiol Ther. 2014 Mar-Apr;37(3):170-9. doi: 10.1016/j.jmpt.2014.02.003. Epub 2014 Mar 15. PMID 24636612
- [Background] Akhtar MW, Karimi H, Gilani SA. Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial. Pak J Med Sci. 2017 Jul-Aug;33(4):1002-1006. doi: 10.12669/pjms.334.12664. PMID 29067082
- [Background] Shamsi MB, Rezaei M, Zamanlou M, Sadeghi M, Pourahmadi MR. Does core stability exercise improve lumbopelvic stability (through endurance tests) more than general exercise in chronic low back pain? A quasi-randomized controlled trial. Physiother Theory Pract. 2016;32(3):171-8. doi: 10.3109/09593985.2015.1117550. Epub 2016 Feb 11. PMID 26864057
- [Background] Ghorbanpour A, Azghani MR, Taghipour M, Salahzadeh Z, Ghaderi F, Oskouei AE. Effects of McGill stabilization exercises and conventional physiotherapy on pain, functional disability and active back range of motion in patients with chronic non-specific low back pain. J Phys Ther Sci. 2018 Apr;30(4):481-485. doi: 10.1589/jpts.30.481. Epub 2018 Apr 13. PMID 29706690
- [Background] Collins JJ, De Luca CJ. The effects of visual input on open-loop and closed-loop postural control mechanisms. Exp Brain Res. 1995;103(1):151-63. doi: 10.1007/BF00241972. PMID 7615030
- [Background] Cano-de-la-Cuerda R, Molero-Sanchez A, Carratala-Tejada M, Alguacil-Diego IM, Molina-Rueda F, Miangolarra-Page JC, Torricelli D. Theories and control models and motor learning: clinical applications in neuro-rehabilitation. Neurologia. 2015 Jan-Feb;30(1):32-41. doi: 10.1016/j.nrl.2011.12.010. Epub 2012 Feb 18. English, Spanish. PMID 22341985
- [Background] Shamsi MB, Sarrafzadeh J, Jamshidi A. Comparing core stability and traditional trunk exercise on chronic low back pain patients using three functional lumbopelvic stability tests. Physiother Theory Pract. 2015 Feb;31(2):89-98. doi: 10.3109/09593985.2014.959144. Epub 2014 Oct 15. PMID 25317504
- [Background] Mousavi SJ, Parnianpour M, Mehdian H, Montazeri A, Mobini B. The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions. Spine (Phila Pa 1976). 2006 Jun 15;31(14):E454-9. doi: 10.1097/01.brs.0000222141.61424.f7. PMID 16778675
- [Background] Rostami M, Noorian N, Mansournia MA, Sharafi E, Babaki AE, Kordi R. Validation of the Persian version of the fear avoidance belief questionnaire in patients with low back pain. J Back Musculoskelet Rehabil. 2014;27(2):213-21. doi: 10.3233/BMR-130439. PMID 24254494
- [Background] Vlaeyen JWS, Seelen HAM, Peters M, de Jong P, Aretz E, Beisiegel E, Weber WEJ. Fear of movement/(re)injury and muscular reactivity in chronic low back pain patients: an experimental investigation. Pain. 1999 Sep;82(3):297-304. doi: 10.1016/S0304-3959(99)00054-8. PMID 10488681
- [Background] Abedi M, Manshadi FD, Khalkhali M, Mousavi SJ, Baghban AA, Montazeri A, Parnianpour M. Translation and validation of the Persian version of the STarT Back Screening Tool in patients with nonspecific low back pain. Man Ther. 2015 Dec;20(6):850-4. doi: 10.1016/j.math.2015.04.006. Epub 2015 Apr 15. PMID 25925506
- [Derived] Raoufi Z, Tabatabaei A, Dadgoo M, Takamjani EE, Salehi R, Sanjari MA. The additional effects of dual-task training with core stability exercises versus general exercises on disability and pain in people with nonspecific chronic low back pain: A randomized controlled trial. Musculoskelet Sci Pract. 2026 Jan 16;82:103501. doi: 10.1016/j.msksp.2026.103501. Online ahead of print. PMID 41633131
- See also: Efficacy of Core Stability in Non-Specific Chronic Low Back Pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8167732/
- See also: Determinants of quality of life in individuals with chronic low back pain: a systematic review — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8741254/
- See also: Chapter 3. European guidelines for the management of acute nonspecific low back pain in primary care — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3454540/
- See also: Effects of attention on the control of locomotion in individuals with chronic low back pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC2387160/
- See also: Compensatory but not anticipatory adjustments are altered in older adults during lateral postural perturbations — https://pubmed.ncbi.nlm.nih.gov/23601702/
- See also: Aging and balance control in response to external perturbations: role of anticipatory and compensatory postural mechanisms — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC4082574/
- See also: Inefficient muscular stabilization of the lumbar spine associated with low back pain. A motor control evaluation of transversus abdominis — https://pubmed.ncbi.nlm.nih.gov/8961451/
- See also: Anticipatory postural control differs between low back pain and pelvic girdle pain patients in the absence of visual feedback — https://pubmed.ncbi.nlm.nih.gov/31726292/
- See also: Changes in motor planning of feedforward postural responses of the trunk muscles in low back pain — https://pubmed.ncbi.nlm.nih.gov/11713638/
- See also: Open-loop and closed-loop postural control mechanisms in Parkinson's disease: increased mediolateral activity during quiet standing — https://pubmed.ncbi.nlm.nih.gov/8552278/
- See also: Open-loop and closed-loop control of posture: a random-walk analysis of center-of-pressure trajectories — https://pubmed.ncbi.nlm.nih.gov/8224055/
- See also: Age-related changes in open-loop and closed-loop postural control mechanisms — https://pubmed.ncbi.nlm.nih.gov/7589299/
- See also: Clinical practice guidelines for the noninvasive management of low back pain: A systematic review by the Ontario Protocol for Traffic Injury Management (OPTIMa) Collaboration — https://pubmed.ncbi.nlm.nih.gov/27712027/
- See also: Which specific modes of exercise training are most effective for treating low back pain? Network meta-analysis — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC7588406/
- See also: Trunk muscle stabilization training plus general exercise versus general exercise only: randomized controlled trial of patients with recurrent low back pain — https://pubmed.ncbi.nlm.nih.gov/15733046/
- See also: Effects of core stabilization exercise and strengthening exercise on proprioception, balance, muscle thickness and pain related outcomes in patients with subacute nonspecific low back pain: a randomized controlled trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC8630919/
- See also: Core Stability Exercise Versus General Exercise for Chronic Low Back Pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5293521/
- See also: Motor Control Exercise for Nonspecific Low Back Pain: A Cochrane Review — https://pubmed.ncbi.nlm.nih.gov/27128390/
- See also: Systematic reviews evaluating the effectiveness of motor control exercises in patients with non-specific low back pain do not consider its principles - A review — https://pubmed.ncbi.nlm.nih.gov/33992272/
- See also: Dual-task interference during initial learning of a new motor task results from competition for the same brain areas — https://pubmed.ncbi.nlm.nih.gov/20434467/
- See also: The Effects of Cognitive Loading on Motor Behavior in Injured Individuals: A Systematic Review — https://pubmed.ncbi.nlm.nih.gov/31066022/
- See also: Effect of dual tasking on anticipatory and compensatory postural adjustments in response to external perturbations in individuals with nonspecific chronic low back pain: Electromyographic analysis — https://pubmed.ncbi.nlm.nih.gov/29332033/
- See also: A meta-analysis of core stability exercise versus general exercise for chronic low back pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC3524111/
- See also: Attention and the control of posture and gait: a review of an emerging area of research — https://pubmed.ncbi.nlm.nih.gov/12127181/
- See also: Effect of dual-tasking on dynamic postural control in individuals with and without nonspecific low back pain — https://pubmed.ncbi.nlm.nih.gov/24636612/
- See also: Effectiveness of core stabilization exercises and routine exercise therapy in management of pain in chronic non-specific low back pain: A randomized controlled clinical trial — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5648929/
- See also: Does core stability exercise improve lumbopelvic stability (through endurance tests) more than general exercise in chronic low back pain? A quasi-randomized controlled trial — https://pubmed.ncbi.nlm.nih.gov/26864057/
- See also: Effects of McGill stabilization exercises and conventional physiotherapy on pain, functional disability and active back range of motion in patients with chronic non-specific low back pain — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC5908986/
- See also: The effects of visual input on open-loop and closed-loop postural control mechanisms — https://pubmed.ncbi.nlm.nih.gov/7615030/
- See also: Theories and control models and motor learning: clinical applications in neuro-rehabilitation — https://pubmed.ncbi.nlm.nih.gov/22341985/
- See also: Comparing core stability and traditional trunk exercise on chronic low back pain patients using three functional lumbopelvic stability tests — https://pubmed.ncbi.nlm.nih.gov/25317504/
- See also: The Oswestry Disability Index, the Roland-Morris Disability Questionnaire, and the Quebec Back Pain Disability Scale: translation and validation studies of the Iranian versions — https://pubmed.ncbi.nlm.nih.gov/16778675/
- See also: Validation of the Persian version of the fear avoidance belief questionnaire in patients with low back pain — https://pubmed.ncbi.nlm.nih.gov/24254494/
- See also: Fear of movement/(re)injury and muscular reactivity in chronic low back pain patients: an experimental investigation — https://pubmed.ncbi.nlm.nih.gov/10488681/
- See also: Translation and validation of the Persian version of the STarT Back Screening Tool in patients with nonspecific low back pain — https://pubmed.ncbi.nlm.nih.gov/25925506/

DOCUMENTS (3):
  • Study Protocol (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05832918/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05832918/SAP_001.pdf
  • Informed Consent Form (2023-03-27): https://cdn.clinicaltrials.gov/large-docs/18/NCT05832918/ICF_003.pdf